CLINICAL TRIAL: NCT05727995
Title: Efficacy of Prophylactic Negative Pressure Wound Therapy (NPWT) on Prevention for Complications After Open Saphenous Vein Harvest in Cardiac Surgery (EFESO Protocol).
Brief Title: Efficacy of Prophylactic Negative Pressure Wound Therapy (NPWT)
Acronym: EFESO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Gianluca Castiello, Principal Investigator, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 126/int/2019
Record Dates: First submitted 2023-02-02; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Wound of Skin
Keywords: negative pressure wound therapy

STUDY DESIGN:
Intervention Model Description: After checking the patients' eligibility they will be blindly randomized in the arm allocation (allocation 1:1).
Who Masked: Outcomes Assessor
Masking Description: The statistician generates the random list and the outcome assessors guarantee the blinding procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The dressing is a polyurethane film with acrylic adhesive that adheres the dressing to the skin surrounding the incision and a polyurethane shell that encapsulates the foam bolster and interface layer, providing a closed system. The PICO pump maintains negative pressure wound therapy (NPWT) at 80mmHg (nominal) +/- 20mmHg to the wound surface. Exudate is managed by the dressing through a combination of absorption and evaporation of moisture through the outer film. PICO is intended for use in wound sizes (surface area x depth) up to 400 cm3, which are considered to be low to moderately exuding. The kit is intended to be used for 7 days on low-exuding wounds and 6 days on moderately exuding wounds. The therapy duration of the kit may be less than indicated if a clinical practice or other factors, such as wound type, wound size, rate or volume of exudate, orientation of the dressing or environmental conditions, result in more frequent dressing changes.
  Interventions: Device: PICO7
- Control group (Sham Comparator): Patients in the control arm will receive a usual care dressing using absorbent cotton pads placed in contact with the wound. Dressings will be applied directly to the wound surface to protect the wound surface environment and the wound bed. Dressing chances are scheduled every 48h.
  Interventions: Other: usual care dressing

INTERVENTIONS:
Device: PICO7 — The use of PICO is contraindicated in the presence of:
  * Patients with malignancy in the wound bed or margins of the wound
  * Previously confirmed and untreated osteomyelitis
  * Nonenteric and unexplored fistulas
  * Necrotic tissue with eschar present
  * Exposed arteries, veins, nerves or organs
  * Exposed anastomotic sites
  * Emergency airway aspiration
  * Pleural, mediastinal or chest tube drainage
  * Surgical suction.
  Arms: Experimental group
Other: usual care dressing — usual care dressing
  Arms: Control group

SUMMARY:
The role of prophylactic negative pressure wound therapy (NPWT) is promising in reducing wound-related complications. However, the prophylactic use of NPWT in reducing wound complications in patients who underwent conventional open harvesting of the great saphenous vein has been under-investigated compering with other surgical approaches.

Therefore, this study aims to assess the effect size of the prophylactic NPWT in preventing wound dehiscence in high-risk patients who underwent conventional open harvesting of the great saphenous vein as a conduit for coronary artery bypass.

DETAILED DESCRIPTION:
The study design is a prospective, randomized, controlled, and monocentric trial. The primary endpoint is given by the reduction of wound dehiscence as a dichotomic outcome (yes versus no).

More precisely, in the experimental group, we will use the proposed device PICO7 (NPWT); this device is certificate CE. PICO consists of a single-use (i.e., completely disposable) NPWT unit, canister, and dressing that are designed for application over clean, closed, sutured, or stapled incisions in a simple peel-and-place process. Instead, in the control group, patients will receive standard care.

Finally, patients eligible to be enrolled in this study will be blindly randomized using for the arm allocation (allocation 1:1). Randomization should take place as soon as possible after consent. Patients will be randomized on a 1:1 basis to receive either dressing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥ 50 years)
* Diagnosis of Diabetes (both type 1 and 2) as comorbidity with anamnesis during the last year of poor glycemic control (HbA1C >7.5%)
* BMI ≥ 25 Kg/m2

Exclusion Criteria:

* Cognitive impairment
* Anamnesis of non-heling wounds
* Wagner grade 2-5 foot wound
* Osteomyelitis
* Pregnancy
* Contraindication to use PICO7 described previously.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Leg wound assessment | At baseline (post-surgery)
  This outcome will be assessed as a categorial variable: a) no complication; b) dehiscence; c) signs of superficial infections. The operative assessment consists of a daily evaluation of the leg wound after the surgery and follow-up assessments.
Leg wound assessment | At 15 days post-surgery
  This outcome will be assessed as a categorial variable: a) no complication; b) dehiscence; c) signs of superficial infections. The operative assessment consists of a daily evaluation of the leg wound after the surgery and follow-up assessments.
Leg wound assessment | At one month post-surgery
  This outcome will be assessed as a categorial variable: a) no complication; b) dehiscence; c) signs of superficial infections. The operative assessment consists of a daily evaluation of the leg wound after the surgery and follow-up assessments.

SECONDARY OUTCOMES:
General in hospital complications | Follow-up 15 days
  General In-hospital clinical complications (yes versus no; if yes, which complications?)
Days of acute hospitalization | Follow-up 30 days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No